CLINICAL TRIAL: NCT05848141
Title: Indoor Rowing as a Novel Exercise Therapy for Cardiovascular Rehabilitation in Middle-Aged and Older Breast Cancer Survivors Following Chemotherapy
Brief Title: Rowing Following Breast Cancer Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202201237
Record Dates: First submitted 2023-03-20; First posted 2023-05-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Survivors
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indoor Rowing (Experimental): Research participants will be instructed how to use a Concept 2 RowErg and will be provided instruction on basic rowing skills for beginners. Exercise training will gradually progress to 50 min of moderate-intensity exercise, on 3 days per week, for 12 weeks.
  Interventions: Behavioral: Exercise training
- Usual Care (No Intervention): Research participants in this group will have the opportunity to complete the supervised indoor rowing program after completing their post-intervention assessments.

INTERVENTIONS:
Behavioral: Exercise training — This is a single site center-based supervised exercise intervention.
  Arms: Indoor Rowing

SUMMARY:
There are more than 3.8 million breast cancer survivors in the United States and cancer survivors have a higher risk of cardiovascular disease (CVD) due to chemotherapy than adults without cancer. Cardiovascular rehabilitation can be an effective strategy to decrease the incidence of CVD and its risk factors in this population. The proposed study may help to examine the effect of a novel exercise intervention on cardiovascular rehabilitation in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary invasive non-metastatic breast cancer, stages I-III
* female based on biological sex
* 40 to 80 years of age
* completed breast cancer treatment 6 to 24 months prior to study enrollment. Adjuvant endocrine therapy for breast cancer (e.g., ovarian suppression, SERMs, SERDs, AIs), CDK4/6 inhibitors, PARP inhibitors, HER2 targeted agents, immunotherapy and bisphosphonates are allowed within 6 months prior to study enrollment and during study participation
* absence of contraindications to exercise or study participation
* study clinician approval

Exclusion Criteria:

* do not meet inclusion criteria
* receiving or scheduled to receive treatment for breast cancer (i.e., chemotherapy, surgery, or radiation) during study participation is not allowed. Adjuvant endocrine therapy, CDK4/6 inhibitors, PARP inhibitors, HER2 targeted agents, immunotherapy and bisphosphonates are allowed during study participation
* lymphedema stage ≥ 2 prior to study enrolment
* any relevant cardiovascular diseases (stroke, heart failure, myocardial ischemia during maximal graded exercise test, myocardial infarction, angina pectoris, coronary artery bypass surgery or angioplasty or coronary stent)
* current participation in other experimental interventions that may confound interpretation of study findings (e.g., dietary intervention for weight loss)
* consistent participation in ≥150 min/week of moderate-intensity rowing exercise training in previous 6 months

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in brachial FMD | Baseline, Following 12 weeks of supervised exercise training
  Flow-mediated dilation (FMD) is an established non-invasive measure of endothelial function. Brachial artery FMD will be determined via ultrasonography in response to reactive hyperemia following 5-min forearm ischemia.
Change in global longitudinal strain | Baseline, Following 12 weeks of supervised exercise training
  Global longitudinal strain is a marker of acute subclinical cardiotoxicity and is recommended for monitoring cancer patients at risk of cancer therapy-related cardiac dysfunction.
% completed vs. planned exercise frequency | Throughout the 12 weeks of supervised exercise training
  We will collect information throughout the exercise intervention regarding % completed vs. planned exercise sessions/week.
% completed vs. planned exercise duration | Throughout the 12 weeks of supervised exercise training
  We will collect information throughout the exercise intervention regarding % completed vs. planned exercise min/session.
% completed vs. planned exercise intensity | Throughout the 12 weeks of supervised exercise training
  We will collect information throughout the exercise intervention regarding % completed vs. planned exercise intensity/session.
Number of participants who experience adverse event as defined by most recent CTCAE | Throughout the 12 weeks of supervised exercise training
  To evaluate safety plans are in place for determination and monitoring of adverse events according to the most recent National Cancer Institute Common Terminology Criteria for Adverse Events. Classification for seriousness, expectedness, severity and relationship to study intervention will be based on the NIH provided definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- Integrative Cardiovasculal Physiology Laboratory, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No